CLINICAL TRIAL: NCT07207135
Title: The Effect of Isometric Exercises Applied to the Quadriceps and Hamstring Muscles at Different Knee Angles on Balance, Joint Position Sense, and Functional Performance in Healthy Individuals
Brief Title: Most Effective Knee Joint Angle Pair for Isometric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Muharrem Gökhan Beydağı, Assistant Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FU_MGBeydagi_Isometric
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Isometric Exercise; Exercise Training; Musculoskeletal Function; Balance, Proprioception, and Functional Performance; Healthy Volunteers
Keywords: Isometric Exercise; Knee Joint Angles; Joint Position Sense; Balance; Functional Performance; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of four parallel groups. Each group performed an eight-week exercise program consisting of progressive resistance training for the hip and ankle combined with isometric quadriceps and hamstring exercises at specific knee joint angles (15°-90°, 30°-105°, 45°-120°, and 60°-135°). The intervention was delivered three times per week under the supervision of physiotherapists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Isometric Exercise at 15° and 90° Knee Angles
  Interventions: Other: Isometric Exercise at 15° and 90° Knee Angles
- Group 2 (Experimental): Isometric Exercise at 30° and 105° Knee Angles
  Interventions: Other: Isometric Exercise at 30° and 105° Knee Angles
- Group 3 (Experimental): Isometric Exercise at 45° and 120° Knee Angles
  Interventions: Other: Isometric Exercise at 45° and 120° Knee Angles
- Group 4 (Experimental): Isometric Exercise at 60° and 135° Knee Angles
  Interventions: Other: Isometric Exercise at 60° and 135° Knee Angles

INTERVENTIONS:
Other: Isometric Exercise at 15° and 90° Knee Angles — Participants performed quadriceps and hamstring isometric contractions at 15° and 90° of knee flexion. Each contraction lasted 10 seconds against resistance, three times per week for eight weeks, with progressive repetitions. Hip and ankle strengthening was also included.
  Arms: Group 1
Other: Isometric Exercise at 30° and 105° Knee Angles — Same protocol as Group 1, but at 30° and 105° of knee flexion.
  Arms: Group 2
Other: Isometric Exercise at 45° and 120° Knee Angles — Same protocol as Group 1, but at 45° and 120° of knee flexion.
  Arms: Group 3
Other: Isometric Exercise at 60° and 135° Knee Angles — Same protocol as Group 1, but at 60° and 135° of knee flexion.
  Arms: Group 4

SUMMARY:
This study investigated the effects of isometric exercises applied to the quadriceps and hamstring muscles at different knee joint angles on balance, joint position sense, and functional performance in healthy individuals. Thirty participants aged 20-30 years were randomized into four groups and performed an eight-week training program, three times per week. Outcome measures included the Y Balance Test, digital goniometer assessments for joint position sense, and functional performance tests (stair climb and 30-second sit-to-stand). The results aim to identify which knee joint angles are most effective for improving neuromuscular function and may guide future rehabilitation and training protocols.

DETAILED DESCRIPTION:
Isometric exercises applied to the quadriceps and hamstring muscles are widely used both in rehabilitation programs and in improving physical fitness in athletes. Isometric contractions occur when the muscle generates tension without changing its length, making them especially suitable in conditions where joint movement is limited or contraindicated. Previous studies have demonstrated the benefits of isometric training in increasing muscle strength, enhancing proprioception, and supporting functional performance. However, there is no clear consensus regarding the effects of isometric exercises performed at different knee joint angles on balance, joint position sense, and functional capacity.

The aim of this study was to investigate the effects of isometric exercises applied to the quadriceps and hamstring muscles at different knee angles (15°-90°, 30°-105°, 45°-120°, 60°-135°) on balance, joint position sense, and functional performance in healthy individuals. Participants aged 20-30 years, without knee pain, previous knee surgery, or pathologies preventing ambulation, were included. All participants were randomized into four groups. Each group performed progressive resistance exercises for the hip and ankle, combined with isometric exercises of the quadriceps and hamstring muscles at the specified knee angles.

The training program lasted eight weeks, with sessions three times per week. During each session, isometric contractions were performed against resistance for 10 seconds at the assigned knee angles, with standardized rest periods between sets. The number of repetitions was progressively increased throughout the program.

Assessments were conducted at baseline and after eight weeks. The following outcome measures were used:

Balance: Y Balance Test

Joint position sense: Digital goniometer measurements

Functional performance: Stair climb test and 30-second sit-to-stand test

The hypothesis of the study was that isometric exercises performed at different knee joint angles would result in different responses in balance, joint position sense, and functional performance. The findings are expected to provide valuable insights both for improving physical fitness in healthy populations and for guiding rehabilitation protocols in clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 30 years
* Voluntary participation with signed informed consent
* No history of knee pain
* No history of knee surgery
* No musculoskeletal pathology preventing ambulation

Exclusion Criteria:

* Presence of cardiovascular or pulmonary diseases that prevent exercise
* Inflammatory or infectious pathology of the knee joint
* Uncontrolled endocrinological disorders or significant systemic/organ insufficiency
* Neurological disorders affecting knee joint innervation

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Balance Performance | Baseline and after 8 weeks of intervention
  Balance will be assessed using the Y Balance Test, which measures dynamic postural control in anterior, posteromedial, and posterolateral directions. Normalized reach distances will be recorded.
Joint Position Sense | Baseline and after 8 weeks of intervention
  Proprioception will be evaluated using a digital goniometer at predetermined knee joint angles (15°, 30°, 45°, 60°, 90°, and 120°). Absolute angular error between target and reproduced angles will be calculated.
Functional Performance- Stair Climb Test | Baseline and after 8 weeks of intervention
  unctional performance will be assessed using the Stair Climb Test (time to ascend and descend 9 steps)

SECONDARY OUTCOMES:
Functional Performance - 30-Second Sit-to-Stand Test | Baseline and after 8 weeks.
  Number of repetitions completed in 30 seconds.

OTHER OUTCOMES:
Sociodemographic and Anthropometric Characteristics | Baseline (prior to intervention)
  aseline demographic and anthropometric variables including age (years), sex (male/female), height (cm), weight (kg), and BMI (kg/m²) will be collected to describe the study population. These measures are not primary or secondary outcomes but will provide descriptive information on participants' characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat Üniversitesi, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No